CLINICAL TRIAL: NCT03049475
Title: Pathophysiology of Acute Pain in Patients With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170056; 17-H-0056
Record Dates: First submitted 2017-02-09; First posted 2017-02-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-04-07

CONDITIONS: Sickle Cell Disease
Keywords: Pain; Cell Free DNA; Inflammatory Markers; Microparticles; NETosis; Natural History
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy, between age 18-80, African/African decent
- Subjects in steady State: Steady state is defined as the period from at any time 8 weeks prior to or after a crisis and samples obtained during this time would be considered steady state samples .

SUMMARY:
Background:

Sickle Cell Disease (SCD) is a blood disorder that occurs mainly in people of African descent. Researchers want to learn more about the painful attacks and complications associated with SCD. They want to look for a relationship between SCD and specific changes in the blood. They want to study the role of genetics, inflammation, and blood clotting factors in SCD. They will do this with blood samples collected during an acute painful attack and in between attacks.

Objective:

To learn more about the painful attacks and complications associated with SCD.

Eligibility:

People ages 18-80 with SCD or who are healthy Africans or African Americans without SCD

Design:

* Participants will be screened with medical history and physical exam.
* Healthy participants will have one visit.
* Participants with SCD will have their first visit when they are not having a pain attack. They will have their next visit during a pain attack. About 3-4 months after this attack, they will have a final visit.
* Visits will include a physical exam, and blood and urine tests.
* Participants may have their blood samples used for genetic testing for research.

DETAILED DESCRIPTION:
Episodic pain is the most common acute morbidity and the leading cause of hospitalization in patients with sickle cell disease. It is caused by microvaso-occlusion induced by sickled red blood cells, an outcome of the polymerization of deoxygenated hemoglobin S (HbS). Factors that contribute to the acute sickle pain include the release of cell-free DNA (cfDNA) and heme that initiate a downstream of events involving inflammation and thrombosis, and ischemia-reperfusion injury.

Cell-free DNA has been shown to be present in plasma of healthy subjects, but elevated in diseases and conditions that are characterized by increased cell death through necrosis or apoptosis. Indeed, we have previously shown that cfDNA in patients with sickle cell disease (SCD) increased dramatically during acute painful episodes. During acute sickle pain, marked elevation of plasma hemoglobin has also been observed due to the acute increase in sickled red blood cells and hemolysis. Both cfDNA and heme (break down product of hemoglobin), act as damage-associated molecular pattern (DAMP) molecules, initiating endothelial inflammation, stimulation of neutrophil extracellular trap (NET) formation, leukocyte recruitment, and microvascular thrombosis.

Although there have been several studies of cytokines and chemokines in steady state and acute sickle cell disease, there has been no comprehensive study of how the inflammatory markers correlate with quantitative levels and profile of cfDNA. In this study, we would like to apply next generation sequencing (NGS) to analyze cfDNA from the plasma of patients with SCD in steadystate, and during painful crises to derive insights on the origin of tissue damage. In parallel with the free plasma DNA, we propose to measure markers of hemolysis and inflammation (cytokines, chemokines), and to investigate if interactions between these circulating molecules and blood cells (e.g. neutrophils) have the potential to modulate the progress and severity of the disease. In addition, we would also like to explore if there is a distinctive cell-free DNA and inflammatory signature in SCD in steady-state and during acute vaso-occlusive crises.

Overall, this study provides an opportunity to evaluate new biomarkers of sickle cell pain crisis and to predict disease severity and prognosis. These measures may allow us to better understand the role of vaso-occlusion, hemolysis, and inflammation-related events and responses and serve as clinical endpoints in future studies of disease pathogenesis and/or therapeutic intervention for sickle cell disease.

ELIGIBILITY:
* SUBJECT INCLUSION CRITERIA (SCD):

  1. Sickle cell disease (all genotypes) with a diagnosis of acute sickle cell pain not related to other cause (if the patient also presents with any other sickle related complication alongside acute sickle pain, including not limited to acute chest syndrome, renal dysfunction, liver dysfunction, stroke and priapism can also be included in the study)
  2. Between 18 and 80 years of age
  3. Ability to provide informed written consent

SUBJECT EXCLUSION CRITERIA (SCD):

1. <18 years of age
2. Pregnancy
3. Chronic inflammatory condition (e.g. SLE, Rheumatoid arthritis or any other infectious process leading to chronic inflammation)
4. Failed stem cell transplantation for SCD
5. On active treatment with cytotoxic or immunosuppressive therapy

INCLUSION CRITERIA FOR HEALTHY CONTROL SUBJECTS:

1. Between 18 and 80 years of age
2. African, of African descent
3. Ability to provide informed written consent

EXCLUSION CRITERIA FOR HEALTHY CONTROL SUBJECTS:

1. Pregnancy
2. Diagnosis of with any of the following chronic disease or conditions:

   1. Sickle cell disease or sickle cell trait
   2. Uncontrolled high blood pressure (systolic blood pressure must not be greater than 160 mmHg or diastolic pressure greater than 90 mmHg
   3. Uncontrolled diabetes (must not have both a documented history of diabetes and random blood glucose of greater than 200 mg/dL)
   4. History of coronary artery disease
   5. History of congestive heart failure
   6. Chronic kidney disease (serum creatinine must not be greater than 2mg/dL)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 subjects with sickle cell disease 40 healthy individuals to serve as controls
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
1. To measure and compare defined sets of markers of obstruction of blood vessels (vaso-occlusion), red cell breakdown (hemolysis), and inflammation during acute painful crisis vs steady state in patients with sickle cell disease. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The team is working on a decision.

REFERENCES:
- [Derived] Tumburu L, Ghosh-Choudhary S, Seifuddin FT, Barbu EA, Yang S, Ahmad MM, Wilkins LHW, Tunc I, Sivakumar I, Nichols JS, Dagur PK, Yang S, Almeida LEF, Quezado ZMN, Combs CA, Lindberg E, Bleck CKE, Zhu J, Shet AS, Chung JH, Pirooznia M, Thein SL. Circulating mitochondrial DNA is a proinflammatory DAMP in sickle cell disease. Blood. 2021 Jun 3;137(22):3116-3126. doi: 10.1182/blood.2020009063. PMID 33661274
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-H-0056.html